CLINICAL TRIAL: NCT00796055
Title: A Phase 1, Open-Label Study of MEDI-547 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Biologic Activity of Intravenous Administration in Subjects With Relapsed or Refractory Solid Tumors Associated With EphA2 Expression
Brief Title: Study of MEDI-547 to Evaluate the Safety, Tolerability, and Biologic Activity of IV Administration in Subjects With Relapsed or Refractory Solid Tumors
Acronym: MEDI-547
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: MI-CP177 study closed per sponsor decision.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP177; NCT00924235 (obsolete NCT alias)
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — MEDI-547

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MEDI-547
  Interventions: Drug: MEDI-547

INTERVENTIONS:
Drug: MEDI-547 — Administered at a dose and schedule as determined by the subject's enrollment cohort as a 60 minute IV infusion as part of a 21-day treatment cycle.

SUMMARY:
To determine the safety, tolerability, and the highest dose of this drug given once every 3 weeks or once every week, (per 21 day cycle) in adult subjects with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
To determine the safety, tolerability, and maximum tolerated dose (MTD) of MEDI 547 in a dose escalation cohort for either administration schedule 1 dose every 3 weeks or 1 dose every week in adult subjects with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For the dose-escalation cohort: cancer relapsed or refractory to at least 1 prior standard care systemic regimen standard therapy with previous histological confirmation of diagnosis of fallopian tube, primary peritoneal, endometrial, cervical, prostate, non-small cell lung, esophageal, gastric, bladder, and renal cell carcinomas or melanoma. Subjects with relapsed or refractory breast, epithelial ovarian, or colon cancer with previous histological confirmation of diagnosis must have progressed through more than 1 prior regimen of therapy. For patients enrolling at the NCI, pathology must be confirmed by the Department of Pathology, CCR, NCI.
* For the dose-expansion cohort: relapsed or refractory epithelial ovarian cancer with progression through more than 1 prior regimen of therapy, or relapsed or refractory fallopian tube, or primary peritoneal cancer with progression after at least 1 prior standard care systemic regimen, with previous histological confirmation of cancer diagnosis. For patients enrolling at the NCI, pathology must be confirmed by the Department of Pathology, Center for Cancer Research (CCR), NCI.
* Patients with the following histologic epithelial ovarian cancer cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (NOS).
* For the dose-expansion cohort of subjects with relapsed or refractory ovarian cancer, subjects must have an archival tumor sample that demonstrates EphA2 expression by immunohistochemical stain.
* Males or females at least 18 years of age at the time of obtaining informed consent.
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to MEDI-547 administration; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy (this is not to include oral or implanted contraceptives (such as the "pill", the "patch", a Depo Provera shot, or hormone laced intrauterine device, but allows the following: non hormonal (copper), intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) beginning at the time the ICF is signed, and must agree to continue using such precautions while receiving MEDI-547 through 30 days after the last dose of MEDI-547.
* For the dose-escalation cohort: measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria is desirable but not required. The following are not considered measurable: pleural effusion or ascites; osteoblastic/osteoclastic lesions or evidence of disease on bone scan alone; progressive irradiated lesions alone, bone marrow involvement, brain metastases, malignant hepatomegaly by physical exam alone; or chemical markers (eg, CA-125, carcinoembryonic antigen [CEA], or prostate specific antigen [PSA]). Recurrent disease following surgery or radiotherapy is measurable provided that 30 days have elapsed since treatment and that measurable disease exists outside the radiation port, or there is clear progression within the radiation port.
* For the dose-expansion cohort: measurable disease, by RECIST criteria is required. The following are not considered measurable: pleural effusion or ascites; osteoblastic/osteoclastic lesions or evidence of disease on bone scan alone; progressive irradiated lesions alone, bone marrow involvement, brain metastases, malignant hepatomegaly by physical exam alone; or chemical markers (eg, CA-125, CEA, or PSA). Recurrent disease following surgery or radiotherapy is measurable provided that 30 days has elapsed since treatment and that measurable disease exists outside the radiation port, or there is clear progression within the radiation port.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Life expectancy of greater than 16 weeks.
* For subjects who had prior treatment with chemotherapy, biological therapy, radiotherapy, or investigational therapy or had prior surgery: eligible for study entry if at least 30 days have passed since their treatment/surgery, provided that all toxicities related to prior treatment have resolved to ≤ Grade 1 severity by National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (NCI CTCAE v3.0 and all surgical wounds have healed.
* Prior immunotherapy with approved agents (eg, trastuzumab, cetuximab, panitumumab, bevacizumab) is allowable if at least 30 days have passed.
* Absolute neutrophil count (ANC) ³ 1500/mm3, platelets ³ 100,000/mm3, hemoglobin > 10.0 g/dL, serum creatinine greater than or equal to 1.5 times the upper limit of normal [ULN] or calculated creatinine clearance > 50 mL/min, serum bilirubin greater than or equal to 2 times the ULN, alkaline phosphatase < 3 times the ULN, and aspartate transferase (AST) and alanine transferase (ALT) greater than or equal to 3 times the ULN.
* Prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR) that are within normal institutional limits.
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization (applies to covered entities in the USA only) obtained from the subject prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Pregnant or lactating women.
* A history of central nervous system metastases or primary central nervous system tumors.
* Symptomatic pleural effusion or ascites requiring paracentesis.
* Symptomatic peripheral neuropathy of Grade 2 or greater.
* Respiratory insufficiency requiring oxygen treatment, or lymphangitic involvement of lungs.
* Any evidence of hematemesis, melena, hematochezia, grade 2 or higher hemoptysis, or gross hematuria. Patients with grade 1 hemoptysis or microscopic hematuria will be permitted on study.
* Active or recent history (within 3 months) of keratitis or conjunctivitis.
* A history of significant adverse events related to a previously administered monoclonal antibody.
* A history of human immunodeficiency virus (HIV) or hepatitis virus infection (HBV,HCV)will be excluded to eliminate the risk of increased adverse events due to immune compromise or liver dysfunction.
* Any evidence or history of myocardial infarction, angina, or arrhythmia (including atrial fibrillation, multifocal premature ventricular contractions, ventricular bigeminy or trigeminy, ventricular tachycardia or requirement for anti-arrhythmics including digoxin), within 6 months prior to initiation of study drug.
* Any evidence of uncontrolled hypertension (systolic blood pressure > 150 mm Hg) within 3 months prior to initiation of investigational product.
* Subjects currently on anticoagulant therapy for thromboembolic disorders or prophylactic reasons will be excluded.
* Any evidence of severe congestive heart failure with severity New York Heart Association classification > Class 1 within the past 12 weeks.
* A marked baseline prolongation of QTc interval (eg, demonstration of QTc interval ≥ 500 millisecs [ms]).
* A prior stroke or transient ischemic attack (TIA) within 6 months prior to initiation of (investigational product) MEDI-547.
* Any evidence of an active infection or systemic use of antimicrobials within 72 hours prior to initial treatment with MEDI-547.
* Current or planned participation (from the day of study entry through 30 days after the last dose of study drug) in a research protocol in which another investigational agent or therapy may be administered.
* Received another investigational agent within 30 days prior to initiation of study drug or not fully recovered from prior investigational treatment.
* A requirement for palliative chemotherapy, hormonal therapy, radiotherapy, surgery, or immunotherapy during the course of the study.
* For subjects in the dose-expansion cohort, history of prior malignancies within the past 5 years other than non-melanomatous skin cancers that have been controlled, carcinoma in situ of the cervix, or superficial bladder cancer.
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
* Any condition that in the opinion of the investigator would interfere with evaluation of the investigational product or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MEDI-547 will be assessed based on the incidence of AEs, SAEs, laboratory abnormalities, physical examination changes, toxicities leading to permanent discontinuation of MEDI-547 and MEDI-547-related deaths. | 30 days after the last dose of MEDI-547.

SECONDARY OUTCOMES:
The antitumor activity of MED-547 will be assessed based on objective response rate (ORR), time to response (TTR), duration of response (DR), time to progression (TTP), progression-free survival (PFS), and overall survival (OS). | 30 days after the last dose of MEDI-547

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Warwick, Study Director — MedImmune LLC
Locations (2):
- United States (2):
  - Research Site, Bethesda, Maryland
  - Research Site, Detroit, Michigan